CLINICAL TRIAL: NCT06606301
Title: Immunohistochemical Expression of EGFR in Oral Squamous Cell Carcinoma- A Cross Sectional Study
Brief Title: Immunohistochemical Expression of EGFR in the Patients Having Oral Squamous Cell Carcinoma
Acronym: EGFR
Status: Completed | Type: Observational
Sponsor: Combined Military Hospital, Pakistan (Other)
Collaborators: National University of Medical Sciences, Pakistan (Other)
Responsible Party: Principal Investigator, Mariya Farooq, M.Phil.Trainee in Oral and Maxillofacial Pathology, Principal Investigator, Combined Military Hospital, Pakistan
Other Study IDs: NUMS/AFPG/21/MPHIL/019
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Oral Cancer , Oral Squamous Cell Carcinoma, Oral Cavity Cancer
Keywords: Oral Squamous Cell Carcinoma, Epidermal Growth Factor Receptor, Marker, Prognosis
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Different Grades of squamous cell carcinoma: Diagnostic test: Biopsy specimens Fresh sections from formalin fixed and paraffin embedded block with sections from the tumor will be prepared followed by Hematoxylin and Eosin staining according to the standard protocol.
  Interventions: Diagnostic Test: BioSB EGFR antibody

INTERVENTIONS:
Diagnostic Test: BioSB EGFR antibody — Appropriate sections from the tumor will be selected basing the choice on tumor content and viability eventually followed by EGFR application which will reveal a brown membrane positivity for the tumor. Total score for RGFR will be calculated by the histopathologists.

SUMMARY:
Oral squamous cell carcinoma (OSCC) is one of the top 10 most common malignancies worldwide. Oral squamous cell carcinoma forms a major health problem in many countries. The reason for the high incidence of oral cavity cancers in Pakistan, and South Asia in general, is the frequent, persistent, and prevalent use of substances classified as oral cancer risk factors. These include betel quid, areca nut, smoking, smokeless tobacco, viral infections such as EBV, HPV, poor oral hygiene (including sharp teeth and decay), ultraviolet (UV) exposure, nutrition, and genetic predisposition.

For several decades the management of OSCC consisted of surgery with or without radiotherapy or chemoradiotherapy. Associated with worse prognosis, overexpression of EGFR may lead to invasion, cellular migration, enhanced angiogenesis, decreased cell apoptosis, and increased metastatic potential. However, advances in immunotherapy have had a major impact on cancer treatment.

This study was exclusively designed to highlight the immunohistochemical detection of expression pattern of EGFR in already diagnosed cases of lip and OSCC in histopathology dept of AFIP and its correlation with the grade of the tumor. In this study, contact details of all diagnosed cases of SCC of lips and oral cavity from June to November 2023 were taken from the archives of Histopathology department. The patients were contacted for consent approval for participation. The data was collected (as per proforma attached), including demographic details, location of tumor. Blocks were retrieved, grade of tumor was identified followed by the application of EGFR marker. Patterns of expression of EGFR were evaluated and compared with grade of tumor to strengthen the correlation of this association.

DETAILED DESCRIPTION:
Oral SCC is a type of cancer that develops from the oral epithelium and accounts for more than 90% of all oral malignancies, with a death rate of more than 140,000 cases globally. It is an invading neoplasm of epithelial origin with various stages of differentiation of squamous cells having a tendency for early and widespread metastatic spread to lymph nodes. It primarily affects individuals in their fifth to sixth decades of life who drink or smoke.

The diagnosis of OSCC requires a combined approach of clinical evaluation, radiological imaging, along with histopathological evaluation. The gold standard for diagnosing OSCC is an incisional/excisional biopsy. Histopathologically, OSCC is characterized by the existence of neoplastic epithelial cells that are invading the underlying connective tissue. The differentiation degree of neoplastic cells determines the histological grade of OSCC, which is an important prognostic factor.

Treatment of OSCC, depending on the current stage of the condition, can be surgery, chemotherapy, radiotherapy, or even a combined approach comprising all these options. Early-stage OSCC can often be cured with surgery or radiotherapy, whereas advanced-stage OSCC has been associated with a worse prognosis.

In conclusion, OSCC is a significant global health issue with an elevated mortality and morbidity in patients with head and neck cancer. Early detection and prompt treatment are crucial in improving the prognosis of OSCC. Oral pathologists and clinicians ought to be mindful of the risk factors, clinical characteristics, and screening requirements for OSCC to ensure timely and accurate diagnosis and treatment for the patients. Targeted therapy has evolved recently as an important treatment modality for cancer, and the most extensively studied pathways for targeted therapy are those related to EGFR.

In the era of personalized medicine, it has been largely accepted that cancer therapy protocols should be devised in light of tumor characteristics of loco-regional population. Previous studies has revealed that the immunohistochemical overexpression of EGFR correlates with poor prognosis. EGFR overexpression is considered an attractive target for anti-EGFR therapy in various tumors. In targeted therapy, entire focus will be on EGFR. This protein has been discovered in 90% of head and neck squamous cell carcinomas. Overexpression of EGFR has unfavorable clinical outcome, poor prognosis and low survival rates in OSCC. To make the diagnosis, clinical correlation with histopathological investigations should be prioritized. There is a strong rationale supporting EGFR-targeting in OSCC. HNSCC is often treated with anti-EGFR antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Cases of surgically treated lip/oral cavity squamous cell carcinoma
* Patients of all age groups, irrespective of their gender
* Patients with a tumor located in the tongue, inferior and superior gingivae, buccal mucosa, floor of the mouth, palate, alveolus and vestibule(buccal/labial and mandible/maxilla)

Exclusion Criteria:

* All specimens with inadequate or poor fixation.
* All specimen of patients having received chemotherapy/radiotherapy prior to surgery
* Very scanty tissue biopsies or those with extensive tissue necrosis
* Patients not consenting to be the part of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the recent biopsy specimens of OSCC submitted to AFIP will be retrieved from the archives of Histopathology department and selected through non probability convenience sampling method.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Correlation of EGFR expression with tumor | 05 months
  To determine the correlation of EGFR with tumor and to establish EGFR as a prognostic marker

SECONDARY OUTCOMES:
Association of EGFR expression with tumor | 05 months
  The EGFR expression was checked for any association with the tumor. A p value of less than 0.05 was taken as significant.

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Farooq, BDS, Principal Investigator — AFIP, Combined Military Hospital
Locations (1):
- Armed Forces Institute of Pathology, Combined Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hashmi AA, Bukhari U, Aslam M, Joiya RS, Kumar R, Malik UA, Zia S, Khan AR, Saleem M, Irfan M. Clinicopathological Parameters and Biomarker Profile in a Cohort of Patients With Head and Neck Squamous Cell Carcinoma (HNSCC). Cureus. 2023 Jul 15;15(7):e41941. doi: 10.7759/cureus.41941. eCollection 2023 Jul. PMID 37588336
- [Background] Gupta S, Pandey P, Verma S, Verma A. p16, p53 and EGFR expression in head and neck squamous cell carcinoma and their correlation with clinicopathological parameters. J Cancer Res Ther. 2024 Apr 1;20(3):881-887. doi: 10.4103/jcrt.JCRT_201_20. Epub 2024 Jun 27. PMID 39023595
- [Background] Bernardes VF, Gleber-Netto FO, Sousa SF, Rocha RM, Aguiar MC. EGFR status in oral squamous cell carcinoma: comparing immunohistochemistry, FISH and CISH detection in a case series study. BMJ Open. 2013 Jan 28;3(1):e002077. doi: 10.1136/bmjopen-2012-002077. PMID 23358562